CLINICAL TRIAL: NCT03176225
Title: Random, Controlled, Single-blinded, Multi-center and Non-inferiority Clinical Study to Evaluate Safety and Effectiveness of XenoSure Biological Patch in the Application of Cardiac Repair
Brief Title: Evaluate Safety and Effectiveness of XenoSure Biological Patch in the Application of Cardiac Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LeMaitre Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P15077-1
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-07

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test Arm (Experimental): In Test Arm, the subjects will be implanted with test article - XenoSure patch. The interventions include: Open heart surgery to address the heart disease; Close the defects with XenoSure Patch
  Interventions: Procedure: Open heart surgery to address the heart disease; Device: Close the defects with XenoSure Patch
- Control Arm (Active Comparator): In Control Arm, the subjects will be implanted with comparator device - Polyester patch by Shanghai Chest Medical Technology Co. The interventions include: Open heart surgery to address the heart disease; Close the defects with Chest Polyester Patch
  Interventions: Procedure: Open heart surgery to address the heart disease; Device: Close the defects with Chest Polyester Patch

INTERVENTIONS:
Procedure: Open heart surgery to address the heart disease — The patient will first have open heart surgery to achieve access to the diseased site in the heart
Device: Close the defects with XenoSure Patch — The heart defects, such as ASD (Atrial Septal Defect) or VSD (Ventricular Septal Defect ), are closed with LeMaitre XenoSure Patch.
  Arms: Test Arm
Device: Close the defects with Chest Polyester Patch — The heart defects, such as ASD (Atrial Septal Defect) or VSD (Ventricular Septal Defect ), are closed with a Polyester Patch made by Shanghai Chest Medical Technology Co.
  Arms: Control Arm

SUMMARY:
The purpose of this clinical trial is to collect safety and effectiveness data to support cardiac repair indication of XenoSure biologic patch. This trial is performed to meet the China FDA regulations for this kind of device. The clinical trial will be performed solely inside China under GCP regulation and all applicable China regulations on medical device clinical trial.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to collect safety and effectiveness data to support cardiac repair indication of XenoSure biologic patch. This trial is performed to meet the China FDA regulations for this kind of device. The clinical trial will be performed solely inside China under GCP regulation and all applicable China regulations on medical device clinical trial.

There will be 144 subjects enrolled, including 72 subjects in the trial arm and 72 subjects in the control arm.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman aged below 6 years old
2. The expected lifetime of no less than 12 months
3. Patients with congenital heart disease in symptoms of ventricular septal defect, atrial septal defect and tetralogy of fallot who need the surgical repair.
4. Physical conditions and vital signs meet requirements for the surgery.
5. The subjects and/or their guardians sign the written Informed Consent Form.

Exclusion Criteria:

1. Patients with severe visceral diseases in liver, kidney, etc.
2. Patients have unstable vital signs and not suitable for the indications.
3. Patients with severe allergic history (especially allergic to bovine materials)
4. Patients with the past medical history of severe immunodeficiency disease
5. The subject has used or plans to use immunomodulatory drugs for more than half a year.
6. The subject with poor blood clotting function, which is defined as that pre-operative INR or APTT is prolonged over 30% than the reference value without drug intervention, or that blood platelet count is less than 100*10^9/L.
7. The subject has severe kidney disorders or diseases with the estimated glomerular filtration rate [GRF]<30mL/min/1.73m2.
8. The subject's ALT or AST level is 2.5 times higher than the upper normal limit or the subject has active liver disease or icterus.
9. The subject has participated in another clinical study within past 3 months or is participating in another clinical study now.
10. The investigator believes that the subject has other reasons unsuitable for inclusion.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Leakage rate at 6 month post-procedure measured by ultrasound | 6 months
  The heart defects should be totally closed by the patch. Any residual flow or leakage, measured by ultrasound, will be recorded. The percentage of the patients that show leakage post-procedure is the failure rate. The study is considered achieved its primary endpoint if the failure rate of the test device is non-inferior to the rate of the comparator device.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No